CLINICAL TRIAL: NCT03122054
Title: Should Surgical Experience Change Our Treatment Strategy on Acute Cholecystitis? Early Versus Delayed Cholecystectomy
Brief Title: Early Versus Delayed Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Canan Tulay ISIL, Ast.Clinical Professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEEAH 12.04.2016/1141
Record Dates: First submitted 2017-03-28; First posted 2017-04-20 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Acute Cholecystitis
Keywords: Laparoscopic Cholecystectomy, Delayed Cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: patients suffering acute pain because of acute cholecystitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (n:88) (Other): patients treated surgically with laparoscopic cholecystectomy immediately
  Interventions: Procedure: laparoscopic cholecystectomy
- Group D (n:88) (Other): patients first treated medically and than treated surgically with delayed (4-8 weeks later) laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — First trocar was inserted with Hasson method (Subumbilical 1 cm vertical incision was made and first 10-mm trocar (VersaportTM plus V2, Covidien, USA) inserted under direct vision) and pneumoperitoneum was created with 12 mm Hg pressure. Second 10-mm trocar was inserted from subxyphoid area. Two 5-mm trocars were inserted in the right upper quadrant area. After general intrabdominal exploration, dissection was started to ensure safe-view of Calot triangle. In case of quite tough gallbladder for griping, gallbladder was drained with a gray intravenous cannula. Cystic artery and cystic duct were separately dissected and twice ligated with Endo Clip™ II ML (Covidien, USA). Gallbladder was dissected from liver bed carefully. Gallbladder was taken out from abdomen through the subumbilical incision.

SUMMARY:
This study examines complications, mortality rates, cost-effectiveness and safety of early laparoscopic cholecystectomy (ELC) versus delayed laparoscopic cholecystectomy (DLC). Group L (n:88) patients treated surgically with laparoscopic cholecystectomy immediately or Group D (n:88) patients first treated medically and than treated surgically with delayed (4-8 weeks later) laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
There is only few knowledge about the comparison of early laparoscopic cholecystectomy (ELC) versus delayed laparoscopic cholecystectomy (DLC) for the treatment of acute cholecystitis considering the surgeon's work experience. This study examines complications, mortality rates, cost-effectiveness and safety of DLC versus ELC. This prospective randomized clinical trial was performed between November 2015-2016 in our General Surgery Clinic. Patients suffering acute cholecystitis in their first 72 hours of pain were enrolled in one of the two study groups: Group L (n:88) patients treated surgically with laparoscopic cholecystectomy immediately or Group D (n:88) patients first treated medically and than treated surgically with delayed (4-8 weeks later) laparoscopic cholecystectomy. All operations and medical treatments were done by surgeons having work experience <2 years.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering acute cholecystitis in their first 72 hours of pain

Exclusion Criteria:

* clinical duration longer than 72 hours, complicated acute cholecystitis (bilirubin >2gr/dl, elevated transaminases (>100 u/l), and cholestatic enzymes (gamma glutamyl transferase >50 u/l), ultrasonographically confirmed dilated intrahepatic or extrahepatic bile ducts, and elevated amylase levels three times more than normal range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Hospital stay | 4 to 8 weeks
  time spent totally in the hospital; time from admission to discharge from hospital in days

SECONDARY OUTCOMES:
Costs of treatment | 4 to 8 weeks
  costs of treatment spent for surgery and hospital stay in days; costs of treatment from admission to discharge from hospital in USD

CONTACTS AND LOCATIONS:
Overall Officials: Riza Gurhan Isil, MD, Principal Investigator — Sağlık Bilimleri Üniversitesi Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi

IPD SHARING:
Plan to Share IPD: No
I can share study data only without sharing patient names and protocol numbers.

REFERENCES:
- [Background] Stinton LM, Shaffer EA. Epidemiology of gallbladder disease: cholelithiasis and cancer. Gut Liver. 2012 Apr;6(2):172-87. doi: 10.5009/gnl.2012.6.2.172. Epub 2012 Apr 17. PMID 22570746
- [Result] Gurusamy K, Samraj K, Gluud C, Wilson E, Davidson BR. Meta-analysis of randomized controlled trials on the safety and effectiveness of early versus delayed laparoscopic cholecystectomy for acute cholecystitis. Br J Surg. 2010 Feb;97(2):141-50. doi: 10.1002/bjs.6870. PMID 20035546